CLINICAL TRIAL: NCT05723003
Title: Multicenter Prospective Validation and Extension of the 'PUMCH' Acute Pulmonary Embolism Severity and Prognosis Prediction Model
Brief Title: Prospective Validation of an Acute Pulmonary Embolism Severity and Prognosis Prediction Model
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCHrule
Record Dates: First submitted 2023-01-09; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; Prognosis assessment model
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to prospectively validate the first PUMCH model for acute PE severity and prognosis prediction based on multi-center data constructed in the pre-project period based on national population data, and to optimize the PUMCH model based on artificial intelligence clustering algorithm.

DETAILED DESCRIPTION:
Patients with pulmonary embolism and aged 18 years or older were enrolled in this study.Patient demographic characteristics(age, sex, department, diagnosis), basic vital signs, symptoms at their admissions (hemoptysis, dyspnea, chest pain, syncope, laboratory examinations (blood lab routines, blood gas, liver and kidney function, myocardial marker), and imaging examinations (vascular ultrasonography, computed tomographic angiography, echocardiography, chest CT,CTPA, pulmonary perfusion imaging, pulmonary angiography, PET/CT) were prospectively collected. Patients were followed up every 1/3/6 months to obtain survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* Inpatients with acute PTE diagnosed by imaging (CTPA, enhanced CT, V/Q imaging suggesting a high probability of PE, pulmonary angiography, MRPA) containing any of the following conditions.

  1. primary acute PTE combined with or without DVT
  2. recurrent acute PTE with a history of previous PTE or DVT
* signed informed consent form

Exclusion Criteria:

* blinded to any diagnostic or therapeutic test (VTE or other conditions)
* unable to complete follow-up (due to cognitive or behavioral limitations, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients with acute PTE diagnosed by imaging (CTPA, enhanced CT, V/Q imaging suggesting a high probability of PE, pulmonary angiography, MRPA).
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | through study completion, an average of 1 year
  all-cause mortality 30 days after diagnosis of acute symptomatic PE.

CONTACTS AND LOCATIONS:
Overall Officials: Juhong Shi, M.D, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China